CLINICAL TRIAL: NCT00937105
Title: Infiltrative Events During Silicone Hydrogel Daily Contact Lens (Daily Wear Corneal Infiltrative Event (DWCIE) Study)
Brief Title: Daily Wear Corneal Infiltrative Event Study
Acronym: DWCIE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Loretta Szczotka-Flynn, OD, PhD, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Results first posted 2014-03-10 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-01

CONDITIONS: Myopia; Hyperopia; Corneal Infiltrative Events
MeSH Terms: conditions — Myopia; Hyperopia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ReNu Multiplus and lotrafilcon A lenses (Active Comparator): ReNu Multiplus contact lens care solution
  Interventions: Device: lotrafilcon A contact lenses; Device: Renu Multiplus
- Clear Care solution and lotrafilcon A lenses (Active Comparator): Clear Care Contact Lens Care Solution
  Interventions: Device: lotrafilcon A contact lenses; Device: Clear Care

INTERVENTIONS:
Device: lotrafilcon A contact lenses — FDA approved soft contact lenses
  Other Names: Air Optix Night & Day Aqua contact lenses
Device: Renu Multiplus
  Arms: ReNu Multiplus and lotrafilcon A lenses
Device: Clear Care
  Arms: Clear Care solution and lotrafilcon A lenses

SUMMARY:
This DWCIE Study is a prospective cohort study of patients fit to the FDA approved and marketed lotrafilcon A (Ciba Vision, Air Optix Night & Day Aqua) soft contact lenses for daily wear (DW) with monthly disposal. 218 healthy myopic (nearsighted) or hyperopic (farsighted) patients with minimal or no astigmatism and no contraindications to DW lens use will be followed for 1 year. The primary outcome is the risk of development of a corneal inflammatory event (CIE) as defined by slit lamp findings and patient symptoms. The main exposure of interest is microbial contamination of study lenses.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be at least 15 years old.
2. The patient must be free of any anterior segment disorders.
3. The patient must have a spectacle corrected spherical refractive error between +5.50 D and -11.00 D with less than or equal to 1.00 D refractive cylinder.
4. The patient must be correctable to 20/25 or better with spectacles.
5. Flat and steep corneal curvatures from Simulated Keratometry readings must be between 39.00 and 48.00 D.
6. Can be successfully fit with lotrafilcon A lenses at the enrollment visit.

Exclusion Criteria

1. The patient has worn rigid gas permeable lenses within the last 30 days or polymethylmethacrylate lenses within the last 3 months.
2. The patient must not be a current successful daily wear user of lotrafilcon A lenses. They may have tried lotrafilcon A lenses in the past, but must not have successfully worn these lenses for daily wear within the last 12 months.
3. The patient has an autoimmune disease (except for Hashimoto's Thyroiditis), immunocompromising disease, connective tissue disease, atopic dermatitis, insulin dependent diabetes, or any other systemic disease that in the investigator's opinion will affect ocular health.
4. The patient is taking chronic systemic medications such as corticosteroids, antimetabolites, or non-steroidal anti-inflammatory agents or any other medication that in the investigator's opinion will affect ocular physiology or study participation.
5. The patient has any ocular disease or condition such as aphakia, corneal dystrophies, corneal edema, external ocular infection, iritis, or had any anterior segment surgery.
6. The patient is taking any ocular medications. If a patient was previously taking any ocular medications, the medications must have been discontinued at least 2 weeks prior to enrollment.
7. The patient must have less than or equal to grade 2 on any of the slit lamp observations of: upper tarsal papilla, corneal staining, corneal neovascularization, conjunctival injection, and lid erythema or scales. Slit lamp findings higher than grade 2 bias the patient toward an adverse event and it may be difficult to detect true change related to contact lens use.
8. The patient is pregnant.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2009-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loretta Szczotka-Flynn, OD, PhD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- Department of Ophthalmology University Hospitals Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Result] Szczotka-Flynn L, Jiang Y, Raghupathy S, Bielefeld RA, Garvey MT, Jacobs MR, Kern J, Debanne SM. Corneal inflammatory events with daily silicone hydrogel lens wear. Optom Vis Sci. 2014 Jan;91(1):3-12. doi: 10.1097/OPX.0000000000000105. PMID 24240354
- [Derived] Jiang Y, Jacobs M, Bajaksouzian S, Foster AN, Debanne SM, Bielefeld R, Garvey M, Raghupathy S, Kern J, Szczotka-Flynn LB. Risk factors for microbial bioburden during daily wear of silicone hydrogel contact lenses. Eye Contact Lens. 2014 May;40(3):148-56. doi: 10.1097/ICL.0000000000000026. PMID 24756119

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From November 2009 to February 2012, 218 participants were randomized at the University Hospitals Case Medical Center Eye Institute.
Pre-assignment Details: Existing soft lens wearers or non contact lens wearers were recruited, no wash out period was required
Period: Overall Study
Arm/Group | Lotrafilcon A Lenses and Clear Care | Lotrafilcon A Lenses and Renu Multiplus
Started | 109 | 109
Completed | 69 | 70
Not Completed | 40 | 39

BASELINE CHARACTERISTICS:
Population: The baseline measures refer to the entire cohort of 218 participants that were randomized, stratified by solution group
Groups:
- Total: Total of all reporting groups
Arm/Group | Lotrafilcon A and Renu | Lotrafilcon A and Clear Care | Total
Number analyzed (Participants) | 109 | 109 | 218
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 3
  Between 18 and 65 years | 108 | 107 | 215
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.4 (11.3) | 34.9 (11.5) | 34.7 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 75 | 153
  Male | 31 | 34 | 65
Region of Enrollment [Number; unit: participants]
  United States | 109 | 109 | 218

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Developing a Corneal Inflammatory Event (CIE)
Description: Raw number of participants in each solution arm developing CIE over 12 month follow-up period
Time Frame: up to 1 year
Population: This primary analysis includes the cohort of all 218 randomized participants. The measured values stratify participants by solution group, however, the statistical analysis reports on the entire cohort (both solution groups) consistent with the primary aim of the study.
Measure: Number; unit: participants
Arm/Group | Lotrafilcon A Lenses and Renu | Lotrafilcon A Lenses and Clear Care
Number analyzed (Participants) | 109 | 109
participants | 6 [88.1 to 96.5] | 7
Statistical Analysis 1: Comparison: Lotrafilcon A Lenses and Renu vs Lotrafilcon A Lenses and Clear Care; Cumulative Unadjusted Probability of Remaining Infiltrate Free in entire Cohort; Test type: Superiority or Other; Kaplan-Meier; Cumulative Unadjusted Probability of remaining CIE-free presented for entire cohort (both solution groups) to remain consistent with the primary aim; Cumulative Probability of no-CIE = 92.8, 95% CI 2-sided [88.6 to 96.9]

2. Secondary Outcome: Number of Participants With CIE Stratified by Microbial Bioburden on Lenses
Description: Microbial bioburden on lenses was determined with predetermined cutoffs to identify substantial bioburden as high levels of normal flora or presence of pathogenic abnormal flora on lenses
Time Frame: up to 1 year
Population: All participants in which valid lens bioburden data was available
Measure: Number; unit: participants
Arm/Group | Participants With Microbial Bioburden on Lenses | Participants Without Microbial Bioburden on Lenses
Number analyzed (Participants) | 53 | 139
participants | 4 [0.490 to 6.156] | 6
Statistical Analysis 1: Comparison: Participants With Microbial Bioburden on Lenses vs Participants Without Microbial Bioburden on Lenses; To determine if microbial contamination of lenses is a risk factor for CIE; Test type: Superiority or Other; p = 0.3923, Regression, Cox; Univariate hazard ratio provided because non-significant finding did not enter into multivariate analyses; Hazard Ratio (HR) = 1.737, 95% CI 2-sided [0.49 to 6.156] — referent is no substantial lens bioburden

3. Secondary Outcome: Number of Participants With CIE Based Stratified by Presence or Absence of Corneal Staining Induced by Solution Use.
Description: Presumed solution induced corneal staining was defined as diffuse punctate fluorescein staining of at least 15% surface area in at least 4 of 5 zones
Time Frame: up to 1 year
Population: Number of participants with valid presumed solution induced corneal staining data in each group
Measure: Number; unit: participants
Arm/Group | Participants With Corneal Staining | Participants Without Corneal Staining
Number analyzed (Participants) | 49 | 145
participants | 2 [0.167 to 10.393] | 8
Statistical Analysis 1: Comparison: Participants With Corneal Staining vs Participants Without Corneal Staining; Test type: Superiority or Other; p = 0.7943, Regression, Cox; Univariate hazard ratio provided because non-significant finding did not enter into multivariate analyses; Hazard Ratio (HR) = 1.316, 95% CI 2-sided [0.167 to 10.393] — referent is no corneal staining

4. Secondary Outcome: Number of Participants With CIE Stratified by Microbial Bioburden on Lens Cases
Description: Microbial bioburden within lens storage cases was determined with predetermined cutoffs to identify substantial bioburden as high levels of normal flora or presence of pathogenic abnormal flora
Time Frame: up to 1 year
Population: All participants in which valid lens case bioburden data was available
Measure: Number; unit: participants
Arm/Group | Participants With Microbial Bioburden on Lens Cases | Participants With no Microbial Bioburden on Lens Cases
Number analyzed (Participants) | 119 | 51
participants | 5 [0.161 to 2.822] | 3
Statistical Analysis 1: Comparison: Participants With Microbial Bioburden on Lens Cases vs Participants With no Microbial Bioburden on Lens Cases; Test type: Superiority or Other; p = 0.5894, Regression, Cox; Univariate hazard ratio provided because non-significant finding did not enter into multivariate analyses; Hazard Ratio (HR) = 0.674, 95% CI 2-sided [0.161 to 2.822] — referent is no substantial case bioburden

5. Secondary Outcome: Number of Participants With CIE Stratified by Overall Microbial Bioburden on Lid Margins
Description: Microbial bioburden on lid margins was determined with predetermined cutoffs to identify substantial bioburden as high levels of normal flora or presence of pathogenic abnormal flora on lids
Time Frame: up to 1 year
Population: All participants in which valid lens bioburden data was available
Measure: Number; unit: participants
Arm/Group | Participants With Microbial Bioburden on Lid Margins | Participants With no Microbial Bioburden on Lid Margins
Number analyzed (Participants) | 154 | 40
participants | 10 [1.10 to 24.70] | 0
Statistical Analysis 1: Comparison: Participants With Microbial Bioburden on Lid Margins vs Participants With no Microbial Bioburden on Lid Margins; Test type: Superiority or Other; p = 0.1742, Regression, Cox — Univariate hazard ratio provided because non-significant finding did not enter into multivariate analyses; Hazard Ratio (HR) = 2.406, 95% CI 2-sided [0.678 to 8.537] — referent is no substantial overall lid bioburden

6. Secondary Outcome: Number of Participants With CIE Stratified by CNS Microbial Bioburden on Lid Margins
Description: Microbial bioburden with coagulase negative staphylococci (CNS) on lid margins was determined with predetermined cutoffs to identify substantial bioburden as high levels of normal CNS flora on lids
Time Frame: up to 1 year
Population: All participants in which valid lids bioburden data was available
Measure: Number; unit: participants
Arm/Group | Participants With CNS Bioburden on Lid Margins | Participants With no CNS Bioburden on Lid Margins
Number analyzed (Participants) | 84 | 110
participants | 8 | 2
Statistical Analysis 1: Comparison: Participants With CNS Bioburden on Lid Margins vs Participants With no CNS Bioburden on Lid Margins; Test type: Superiority or Other; p = 0.04, Regression, Cox; Multivariate model adjusted for solution, gender and age; Hazard Ratio (HR) = 5.22, 95% CI 2-sided [1.10 to 24.70] — referent is no substantial CNS lid bioburden

ADVERSE EVENTS:
Time Frame: up to 1 year
Description: CIE definitions adopted from the standards as listed in the "Institute for Eye Research/L.V. Prasad Eye Institute (IER/LVPEI) Guide To Corneal Infiltrative Conditions
  Contact Lens Papillary Conjunctivitis was a clinical diagnosis that required temporary or permanent discontinuation of lens wear due to large papilla upon upper lid eversion
Arm/Group | Entire Cohort of Lotrafilcon A Users
Serious Adverse Events (participants affected / at risk) | 1/218
Other Adverse Events (participants affected / at risk) | 23/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Entire Cohort of Lotrafilcon A Users (N=218)
microbial keratitis (Eye disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Entire Cohort of Lotrafilcon A Users (N=218)
corneal infiltrative event (Eye disorders) | 12
Contact Lens Papillary Conjunctivitis (Eye disorders) | 11

LIMITATIONS AND CAVEATS:
Mostly asymptomatic CIE events occurred which limited the ability to retrieve the lens worn (for culture) precisely at the time of CIE development; this may have hindered our ability to capture bioburden at the time of the adverse event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less